CLINICAL TRIAL: NCT06995950
Title: Legume Allergy in Children: Improving Diagnosis Through the Development of Molecular Allergy Testing
Brief Title: Improving Diagnosis of Legume Allergy in Children
Acronym: LACID
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Principal Investigator, Amandine DIVARET-CHAUVEAU, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI140
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Food Allergy in Children; Legumes Allergy; Molecular Diagnostic
Keywords: food allergy; legume; children; molecular allergology
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, almost 15% of serious food allergies in children are caused by legumes, especially peanuts. Other legumes like soy, lentils, peas, lupin, chickpeas, beans, and fenugreek can also cause allergic reactions.

But here's the problem: only peanuts, soy, and lupin are required to be clearly labeled on food packaging in the European Union. This makes it hard for families to know when other legumes-like peas or fenugreek-are hidden in processed foods.

Avoiding all these legumes is hard-especially since many of them are used in processed foods and not always listed on the label. Right now, detailed allergy tests to evaluate the probability of allergy diagnosis are only available for peanuts and soy, and not for other legumes.

LACID study has been created to find and study the proteins in lupin, fenugreek, and peas that may cause allergies and developp better allergy tests for these legumes-possibly as part of a diagnostic tool that can give clear results using just a blood sample.

The goal is to help doctors and families better understand which legumes a child really needs to avoid-and which ones are actually safe to eat.

DETAILED DESCRIPTION:
In France, almost 15% of serious food allergies in children are caused by legumes, especially peanuts. Other legumes like soy, lentils, peas, lupin, chickpeas, beans, and fenugreek can also cause allergic reactions.

But here's the problem: only peanuts, soy, and lupin are required to be clearly labeled on food packaging in the European Union. This makes it hard for families to know when other legumes-like peas or fenugreek-are hidden in processed foods.

At the same time, legumes are being used more and more. They are healthy, rich in protein, and better for the environment. In France, a 2019 law (called EGALIM) requires at least one vegetarian meal per week in schools, and these meals often use legumes to replace meat. To make them more appealing to kids, legumes are turned into foods that look familiar-like veggie nuggets or burgers. As a result, children are eating more legumes, often without knowing it.

Children who are allergic to peanuts are often also sensitised to other legumes. This is because the proteins in different legumes can be similar. But being "sensitised" doesn't mean a child will have a real allergic reaction when eating that food.

Previously, a retrospective study conducted in Nancy, France, looked at nearly 200 children allergic to peanuts. In this study, 2 out of 3 children were sensitised to at least one other legume, 1 out of 5 was truly allergic to another legume and allergy was confirmed in 16% of cases for fenugreek, 56% for lupin, and 45% for peas.

Avoiding all these legumes is hard-especially since many of them are used in processed foods and not always listed on the label. Lupin can be hidden in pastries, fenugreek is found in spice mixes and even some cheeses or medicines and peas are used in vegetarian dishes like veggie steaks or nuggets.

This makes everyday life stressful for allergic children and their families. Right now, the only sure way to know if a child is allergic to a food is to do a carefully supervised food oral challenge at the hospital. But scientists are trying to find easier, safer ways to diagnose legume allergies-so that children don't have to avoid foods unnecessarily.

So far, detailed allergy tests are available for peanuts and soy, but not for other legumes. LACID study has been created to find and study the proteins in lupin, fenugreek, and peas that may cause allergies and developp better allergy tests for these legumes-possibly as part of a diagnostic tool that can give clear results using just a blood sample.

The goal is to help doctors and families better understand which legumes a child really needs to avoid-and which ones are actually safe to eat.

ELIGIBILITY:
Inclusion Criteria:

* Sensitised to lupine, fenugreek or pea

Exclusion Criteria:

* on going anti-IgE treatment or in the last 6 months

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children sensitised to lupine, fenugreek or pea, treated in French Allergy Pediatric units, with data regarding tolerance of at least one these three legumes
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Legume allergy | in the past 2 years before recruitment and until the end of recruitment
  Number of children with a confirmed allergy to pea, fenugreek or lupin (an allergic reaction in real life or a positive oral food challenge)

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Divaret-Chauveau, MD, PhD, Principal Investigator — Pediatric Allergy Unit, University Hospital of Nancy

IPD SHARING:
Plan to Share IPD: Undecided